CLINICAL TRIAL: NCT03846557
Title: PRospective Evaluation Complementing Investigation With Acurate Neo Device
Acronym: PRECISA
Status: Completed | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: PRECISA -EPIC 11
Record Dates: First submitted 2019-02-11; First posted 2019-02-19 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2022-01

CONDITIONS: Aortic Stenosis
Keywords: TAVI; Valve
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Treatment: Transcatheter Aortic Valve Implantation (TAVI) Device
  Interventions: Device: Transcatheter Aortic Valve Implantation (TAVI)

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation (TAVI) — Implantation of the Acurate Neo Transcatheter Heart Valve

SUMMARY:
The study collects real-world data of patients who were treated with the Acurate Neo TAVI System and evaluates early and midterm clinical outcomes.

DETAILED DESCRIPTION:
The study collects real-world data of patients who were treated with the Acurate Neo TAVI System and evaluates early and midterm clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years.
* Severe aortic stenosis with indication of implantation of aortic valve prosthesis in which an Acurate Neo device is implanted according to the indications for use.
* Has signed the Patient Informed Consent Form.

Exclusion Criteria:

* Severe aortic stenosis without indication of implantation of aortic valve prosthesis in which an Acurate Neo device is implanted according to the indications for use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe aortic stenosis with indication of implantation of aortic valve prosthesis in which an Acurate Neo device is implanted according to the indications for use.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
Device success of implantation | 7 days
  Proportion of patients with device success of implantation defined as:
  * absence of procedural mortality AND
  * correct positioning of a single prosthetic heart valve into the proper anatomical location AND
  * no prosthesis - patient mismatch AND
  * mean aortic valve gradient <20 mmHg, AND
  * no moderate or severe prosthetic valve regurgitation
Cardiovascular death | 30 days post-index procedure
  Cumulative incidence of a combination of all cause Cardiovascular death

SECONDARY OUTCOMES:
Assessment of early safety | 30 days
  Proportion of patients with early safety defined by the Valve Academic Research Consortium-2 (VARC-2) as:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Life-threatening bleeding
  * Acute kidney injury-Stage 2 or 3 (including renal replacement therapy)
  * Coronary artery obstruction requiring intervention
  * Major vascular complication
  * Valve-related dysfunction requiring repeat procedure
Assessment of time-related valve safety | 30 days
  Proportion of patients with structural valve deterioration as defined by:
  * Requiring repeat procedure (transcatheter or surgical heart valve replacement)
  * Valve-related dysfunction defined by
    * mean aortic valve gradient ≥20 mmHg and
    * no moderate or severe prosthetic valve regurgitation
  * Prosthetic valve endocarditis
  * Prosthetic valve thrombosis
  * Thrombo-embolic events (e.g. stroke)
  * VARC bleeding, unless clearly unrelated to valve therapy
Assesment of NYHA (New York Heart Association ) classification | 7 days, 30 days, 12 month
  Assesment of NYHA classification
Assessment of mean aortic gradient post-implantation | up to one year
  Assessment of mean aortic gradient post-implantation
Death during the hospitalization of the patient | date of procedure till date of estimated discharge, assessed up to two weeks
  Proportion of patients with death during the hospitalization designated by the VARC-2 criteria

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Hospital Universitari Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Clinico de San Carlos, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital Universitari I Politècnic de La Fé, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Background] Adams DH, Popma JJ, Reardon MJ. Transcatheter aortic-valve replacement with a self-expanding prosthesis. N Engl J Med. 2014 Sep 4;371(10):967-8. doi: 10.1056/NEJMc1408396. No abstract available. PMID 25184874
- [Background] Leon MB, Smith CR, Mack MJ, Makkar RR, Svensson LG, Kodali SK, Thourani VH, Tuzcu EM, Miller DC, Herrmann HC, Doshi D, Cohen DJ, Pichard AD, Kapadia S, Dewey T, Babaliaros V, Szeto WY, Williams MR, Kereiakes D, Zajarias A, Greason KL, Whisenant BK, Hodson RW, Moses JW, Trento A, Brown DL, Fearon WF, Pibarot P, Hahn RT, Jaber WA, Anderson WN, Alu MC, Webb JG; PARTNER 2 Investigators. Transcatheter or Surgical Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2016 Apr 28;374(17):1609-20. doi: 10.1056/NEJMoa1514616. Epub 2016 Apr 2. PMID 27040324
- [Background] Reardon MJ, Van Mieghem NM, Popma JJ, Kleiman NS, Sondergaard L, Mumtaz M, Adams DH, Deeb GM, Maini B, Gada H, Chetcuti S, Gleason T, Heiser J, Lange R, Merhi W, Oh JK, Olsen PS, Piazza N, Williams M, Windecker S, Yakubov SJ, Grube E, Makkar R, Lee JS, Conte J, Vang E, Nguyen H, Chang Y, Mugglin AS, Serruys PW, Kappetein AP; SURTAVI Investigators. Surgical or Transcatheter Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2017 Apr 6;376(14):1321-1331. doi: 10.1056/NEJMoa1700456. Epub 2017 Mar 17. PMID 28304219
- [Background] Thyregod HG, Steinbruchel DA, Ihlemann N, Nissen H, Kjeldsen BJ, Petursson P, Chang Y, Franzen OW, Engstrom T, Clemmensen P, Hansen PB, Andersen LW, Olsen PS, Sondergaard L. Transcatheter Versus Surgical Aortic Valve Replacement in Patients With Severe Aortic Valve Stenosis: 1-Year Results From the All-Comers NOTION Randomized Clinical Trial. J Am Coll Cardiol. 2015 May 26;65(20):2184-94. doi: 10.1016/j.jacc.2015.03.014. Epub 2015 Mar 15. PMID 25787196
- [Background] Baumgartner H, Falk V, Bax JJ, De Bonis M, Hamm C, Holm PJ, Iung B, Lancellotti P, Lansac E, Rodriguez Munoz D, Rosenhek R, Sjogren J, Tornos Mas P, Vahanian A, Walther T, Wendler O, Windecker S, Zamorano JL; ESC Scientific Document Group. 2017 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2017 Sep 21;38(36):2739-2791. doi: 10.1093/eurheartj/ehx391. No abstract available. PMID 28886619
- [Background] Iung B, Baron G, Butchart EG, Delahaye F, Gohlke-Barwolf C, Levang OW, Tornos P, Vanoverschelde JL, Vermeer F, Boersma E, Ravaud P, Vahanian A. A prospective survey of patients with valvular heart disease in Europe: The Euro Heart Survey on Valvular Heart Disease. Eur Heart J. 2003 Jul;24(13):1231-43. doi: 10.1016/s0195-668x(03)00201-x. PMID 12831818
- [Background] Pesarini G, Lunardi M, Piccoli A, Gottin L, Prati D, Ferrero V, Scarsini R, Milano A, Forni A, Faggian G, Ribichini F. Effectiveness and Safety of Transcatheter Aortic Valve Implantation in Patients With Pure Aortic Regurgitation and Advanced Heart Failure. Am J Cardiol. 2018 Mar 1;121(5):642-648. doi: 10.1016/j.amjcard.2017.11.042. Epub 2017 Dec 11. PMID 29329825
- [Derived] Tebar D, Carrillo X, Garcia Del Blanco B, Gomez-Hospital JA, Nombela L, Molina E, Galeote G, Vilalta V, Serra-Garcia V, Carol GM, Jimenez-Valero S, Fernandez-Nofrerias E, Calabuig-Goena A, Jurado-Roman A, Sanchez-Recalde A, Velasco MF, Bosca L, Moreno R. Experience with the ACURATE neo and neo2 transcatheter aortic valves in Spain. The PRECISA (PRospective Evaluation Complementing Investigation with ACURATE devices) registry. Catheter Cardiovasc Interv. 2024 May;103(6):1015-1022. doi: 10.1002/ccd.31032. Epub 2024 Apr 5. PMID 38577931